CLINICAL TRIAL: NCT07388069
Title: A Proof of Concept, Open-label, Two-arm Study to Investigate the Safety and Preliminary Efficacy of TN-001 Topical Eyedrops in Male and Female Patients With Progressive Keratoconus.
Brief Title: Study of TN-001 Topical Eyedrops for Keratoconus
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TheiaNova Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TN-001-01
Record Dates: First submitted 2026-01-15; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Keratoconus
Keywords: keratoconus; eyedrops; non-invasive; Transforming Growth Factor
MeSH Terms: conditions — Keratoconus | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: This is a two-arm study investigating a low and a high dose of TN-001. A total of 20 participants will be enrolled (ten in each arm).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose (Experimental): Low dose TGF-B3 and Dexamethasone Sodium Phosphate
  Interventions: Drug: Low-dose TGF-B3 and Dexamethasone Sodium Phosphate
- High-dose (Experimental): High dose TGF-B3 and Dexamethasone Sodium Phosphate
  Interventions: Drug: High-dose TGF-B3 and Dexamethasone Sodium Phosphate

INTERVENTIONS:
Drug: Low-dose TGF-B3 and Dexamethasone Sodium Phosphate — Low-dose TGF-B3 and Dexamethasone Sodium Phosphate
  Arms: Low-dose
Drug: High-dose TGF-B3 and Dexamethasone Sodium Phosphate — High-dose TGF-B3 and Dexamethasone Sodium Phosphate
  Arms: High-dose

SUMMARY:
The goal of this clinical trial is to learn if TN-001, a new eye-drop therapy, is safe and well-tolerated in adult patients with progressive keratoconus. It will also provide data on whether this therapy is effective in treating keratoconus.

The main questions it aims to answer are:

What medical problems do participants have when using TN-001 eyedrops? Does TN-001 eyedrop therapy stop keratoconus from progressing further?

Participants will:

Take TN-001 eyedrops twice a day, every day, for 3-6 weeks. Visit the clinic once every week for checkups and tests. Keep a diary of their symptoms.

DETAILED DESCRIPTION:
TN-001, the study drug, is a topical eyedrop containing Transforming Growth Factor Beta 3 (TGFB3) and Dexamethasone Sodium Phosphate (DexSP). It is anticipated that TN-001 may produce collagen in the eye, which is believed to stiffen the cornea. Stiffening of the cornea is desirable in patients with keratoconus as it helps to stop disease progression.

The purpose of this study is to:

* Evaluate the safety of TN-001
* Evaluate whether TN-001 eye drops are well tolerated in and around the eye
* Provide an initial indication on whether TN-001 may be effective in treating progressive keratoconus.
* Provide an indication of the duration of treatment impact.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 to 40 years of age inclusive, at the time of signing the informed consent.
2. Diagnosed with progressive keratoconus in one or both eyes.
3. Minimum corneal thickness equal to or greater than 400 microns.
4. Maximum corneal keratometry of 45 D to 54 D.
5. Willing and able to comply with all clinic visits and study-related procedures and instructions.
6. Able to self-medicate or be assisted with applying study eye drops twice daily for trial duration.
7. Provide signed informed consent to participate in the study.

Exclusion Criteria:

1. Concurrent use of contact lenses, including rigid gas permeable lenses
2. Known allergy to steroids, growth factors or gellan gum
3. Presence of ocular surface inflammation at any screening visit
4. Recurrent corneal erosions
5. Significant central corneal scarring or hydrops
6. Previous corneal cross-linking
7. Previous corneal transplant
8. Previous corneal or intraocular surgeries
9. Presence of any other ocular disease of the eye (not limited to cornea) e.g. glaucoma, uveitis, uncontrolled diabetic retinopathy
10. Presence or history of ocular cancer
11. Prior ocular trauma or prior retinal detachment involving the macula
12. Received an ocular corticosteroid within the past 6 months (within the past 3 months, for topical ocular corticosteroids), or any intravitreal injection within the last 6 months in the study eye prior to day 0
13. Any severe comorbid condition or other issue that renders the participant unsuitable for participation in the study
14. A comorbid condition with an estimated life expectancy of ≤6 months at the time of consent
15. Systemic comorbidities that pose a significant surgical risk
16. Current use or anticipated use during the study of a systemic corticosteroid with a dose greater than 10mg daily, or an immunosuppressant agent by any route (oral, injectable)
17. Current use or anticipated use during the study of medicated lubricating eye drops or topical ophthalmic antihistamines
18. History of connective tissue disorders, collagenoses, collagen vascular diseases, autoimmune or other immune deficiency disease
19. Pregnancy or planning to become pregnant
20. Participation in another interventional clinical trial within 30 days or 5 half-lives of that Investigational Product prior to consent for this trial, or planning to participate in another clinical trial at the time of consent
21. Known alcohol, drug or medication abuse within 1 year prior to consent for this study
22. Treatment with an anticancer therapy (chemotherapy, immunotherapy, radiotherapy, targeted therapy or gene therapy) within 3 months prior to day 0 or at any time during the study. Recovery from any associated toxicities must be documented prior to inclusion
23. Mental condition rendering the participant unable to understand the nature, scope, and possible consequences of the study
24. Participants who are employees of the Sponsor, study site or their immediate families
25. Inability or unwillingness to comply with all follow-up through to the end of the study, and/or unwilling to allow access to review medical records in accordance with local regulatory requirements at the time of consent
26. Retinal disease, including proliferative diabetic retinopathy, retinal fibrosis, neovascular age-related macular degeneration
27. Participants in whom corneal thinning has stabilized by ophthalmologist's opinion during screening
28. Myopic degeneration with potential acuity less than 20/40 in either eye
29. Any reason for which in the opinion of the principal investigator the participant should not be enrolled into the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Participant-reported ocular tolerability score (5-point scale) | Baseline (Day 1) to Day 180 of treatment initiation
  Participant-reported ocular tolerability was assessed using a study-specific eye questionnaire measured on a 5-point ordinal scale in the treatment eye.
Incidence of ocular and peri-ocular inflammation by slit-lamp examination | Baseline (Day 1) through Day 180
  Incidence of inflammation of the eye and surrounding tissues, including redness, aqueous cells, flare, limbus, fornices, tear ducts, and meibomian glands, assessed by slit-lamp microscopy using the Efron scale or a similar numerical grading scale in the treatment eye.
Incidence of corneal scarring and conjunctival inflammation | Baseline (Day 1) through Day 180
  Incidence of corneal scarring and conjunctival inflammation assessed by slit-lamp microscopy using the Efron scale or a similar numerical grading scale in the treatment eye.
Increase from baseline in intraocular pressure (mmHg) | Baseline (Day 1) through Day 180
  Increase from baseline in intraocular pressure measured using a hand-held tonometer (mmHg) in the treatment eye.
Change from baseline in endothelial cell count (cells/mm²) | Baseline (Day 1) through Day 180
  Change from baseline in endothelial cell count measured using specular microscopy (cells/mm²) in the treatment eye.
Change from baseline in endothelial cell characteristics | Baseline (Day 1) through Day 180
  Change from baseline in endothelial cell characteristics, including coefficient of variation and percentage of hexagonal cells, measured using specular microscopy in the treatment eye.
Incidence of structural corneal and ocular surface changes | Baseline (Day 1) through Day 180
  Incidence of structural changes of the cornea and ocular surface, including corneal opacities, corneal haze, and keratitis, assessed by anterior segment optical coherence tomography in the treatment eye.
Change from baseline in stromal thickness (microns) | Baseline (Day 1) through Day 180
  Change from baseline in stromal thickness measured in microns using anterior segment optical coherence tomography in the treatment eye.
Change from baseline in choroidal and retinal thickness | Baseline (Day 1) through Day 180
  Change from baseline in choroidal and retinal thickness measured using optical coherence tomography in the treatment eye.
Incidence of abnormal findings on dilated fundus examination | Baseline (Day 1) through Day 180
  Incidence of pathology involving the retina, optic nerve, lens, and/or macula assessed by dilated fundus examination using slit-lamp microscopy with a fundus lens in the treatment eye.
Change from baseline in visual acuity (LogMAR) | Baseline (Day 1) through Day 180
  Change from baseline in visual acuity measured using a LogMAR chart in the treatment eye.

SECONDARY OUTCOMES:
Change from baseline in corneal stiffness and biomechanics | Baseline (Day 1) to Day 180 of treatment initiation
  Change from baseline in corneal stiffness and biomechanical parameters measured using the Oculus Corvis® ST in the treatment eye.
Change from baseline in maximum corneal curvature (Kmax) | Baseline (Day 1) through Day 180
  Change from baseline in maximum corneal curvature measured using central keratometry (Kmax) with the Oculus Pentacam in the treatment eye.
Change from baseline in mean central corneal curvature | Baseline (Day 1) through Day 180
  Change from baseline in mean central corneal curvature measured using keratometry with the Oculus Pentacam in the treatment eye.
Change from baseline in corneal thickness (pachymetry) | Baseline (Day 1) through Day 180
  Change from baseline in corneal thickness (pachymetry), measured in microns using the Oculus Pentacam in the treatment eye.
Change from baseline in corneal shape (Belin ABCD parameters) | Baseline (Day 1) through Day 180
  Change from baseline in corneal shape assessed using Belin ABCD parameters measured with the Oculus Pentacam in the treatment eye.
Change from baseline in corneal higher-order aberrations | Baseline (Day 1) through Day 180
  Change from baseline in corneal higher-order aberrations, including spherical and coma-like aberrations, measured using Pentacam wavefront aberrometry in the treatment eye.

OTHER OUTCOMES:
Change from baseline in ocular stiffness parameters measured by Oculus Corvis® ST | Baseline (Day 1) to Day 180 of treatment initiation
  Change from baseline in ocular stiffness parameters in participants with keratoconus, measured using the Oculus Corvis® ST in the treatment eye, to evaluate persistence of biomechanical changes through Day 180. The specific parameters assessed include:
  * Stiffness Parameter at First Applanation (SP-A1, N/m)
  * Stiffness Parameter at Highest Concavity (SP-HC, N/m)
  * Deformation Amplitude Ratio at 2 mm (DA Ratio 2 mm, ratio)
  * Integrated Inverse Radius (m-¹)
  * Stress-Strain Index (SSI, range 0-1)
Change from baseline in corneal parameters associated with disease progression in the treatment eye | Baseline (Day 1) to Day 180 of treatment initiation
  Change from baseline in corneal parameters associated with disease progression in the treatment eye in participants with keratoconus, evaluated through Day 180. The specific measurements assessed include:
  Corneal curvature (keratometry):
  * Maximum keratometry (Kmax, diopters)
  * Zonal maximum keratometry (Zonal Kmax, diopters)
  Corneal thickness (pachymetry):
  - Corneal thickness (microns)
  Corneal shape (topography):
  - Belin ABCD classification parameters (continuous measures)
  Corneal aberrations:
  * Root Mean Square (RMS) total aberrations (µm)
  * RMS low-order aberrations (LOA, µm)
  * RMS high-order aberrations (HOA, µm)
  * HOA spherical aberration (µm)
  * HOA coma aberration (µm)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Trials Australia, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Diekman BO, Rowland CR, Lennon DP, Caplan AI, Guilak F. Chondrogenesis of adult stem cells from adipose tissue and bone marrow: induction by growth factors and cartilage-derived matrix. Tissue Eng Part A. 2010 Feb;16(2):523-33. doi: 10.1089/ten.TEA.2009.0398. PMID 19715387
- [Background] CULLEN JF, BUTLER HG. MONGOLISM (DOWN'S SYNDROME) AND KERATOCONUS. Br J Ophthalmol. 1963 Jun;47(6):321-30. doi: 10.1136/bjo.47.6.321. No abstract available. PMID 14189698
- [Background] Carrington LM, Albon J, Anderson I, Kamma C, Boulton M. Differential regulation of key stages in early corneal wound healing by TGF-beta isoforms and their inhibitors. Invest Ophthalmol Vis Sci. 2006 May;47(5):1886-94. doi: 10.1167/iovs.05-0635. PMID 16638995
- [Background] Bawazeer AM, Hodge WG, Lorimer B. Atopy and keratoconus: a multivariate analysis. Br J Ophthalmol. 2000 Aug;84(8):834-6. doi: 10.1136/bjo.84.8.834. PMID 10906086
- [Background] Ambekar R, Toussaint KC Jr, Wagoner Johnson A. The effect of keratoconus on the structural, mechanical, and optical properties of the cornea. J Mech Behav Biomed Mater. 2011 Apr;4(3):223-36. doi: 10.1016/j.jmbbm.2010.09.014. Epub 2010 Oct 7. PMID 21316609